CLINICAL TRIAL: NCT01391416
Title: Prevalence Of Hyperhomocysteinemia In Thai CKD Patients And Relationship To Cardiovascular Events: Subgroup Analysis From Thai SEEK Study
Brief Title: Prevalence Of Hyperhomocysteinemia In Thai Chronic Kidney Disease (CKD) Patients
Status: Completed | Type: Observational
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Thananda Trakarnvanich, Renal Unit,Department of Medicine,Faculty of Medicine,Vajira Hospital
Other Study IDs: VJR-0002
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2010-05

CONDITIONS: Cardiovascular Disease; Hyperhomocysteinemia
Keywords: Hyperhomocysteinemia; Chronic kidney disease
MeSH Terms: conditions — Cardiovascular Diseases; Hyperhomocysteinemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CKD stage 3-4: CKD stage 3-4 from Thai SEEK study
- hyperhomocysteine group: CKD stage 3-4 from Thai SEEK study

SUMMARY:
It is well recognized that patients with chronic kidney disease (CKD) have an increased risk for cardiovascular disease (CVD) and hyperhomocysteinemia appears to be a predictor of future CVD events. Hyperhomocysteinemia has been reported to bo of high prevalence in patients with CKD. The investigators aim to study the prevalence of hyperhomocysteinemia in Thai CKD patients by using Thai Screening and Early Evaluation of Kidney Disease (SEEK) study database and their relationship to CVD.

DETAILED DESCRIPTION:
Ninety eight subjects were sampling from Thai SEEK study database Traditional Traditional risk factors of CVD such as total cholesterol, triglyceride, age, sex, history of smoking and blood pressure levels were examined and recorded. Stored sera of these subjects were analyzed for the total homocysteine (tHcy) level. Analysis of variance was used to evaluate the different of mean tHcy among groups

ELIGIBILITY:
Inclusion Criteria:

* CKD stages 3-4 from Thai SEEK Study

Exclusion Criteria:

* CKD stage 5

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ninety eight subjects from CKD stages 3-4 were randomly sampling from Thai- SEEK study database. Thai-SEEK study is a community-based cross-sectional survey that was conducted between August 2007-june 2008 in four regions of Thailand (i.e Northern, Northeastern, Central and Southern) and Bangkok (Metropolitan).
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Level of Homocysteine | 3 months
  Level of homocysteinemia according to each CKD level

SECONDARY OUTCOMES:
Association of cardiovascular event to the level of homocysteine | 3 months
  Hugh level of homocysteine will have association with cardiovascular events or not

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, M.D., Principal Investigator — Renal Unit,Department of Medicine,Faculty of Medicine,Vajira Hospital,University of Bangkok Metropolis

REFERENCES:
- [Background] Ingsathit A, Thakkinstian A, Chaiprasert A, Sangthawan P, Gojaseni P, Kiattisunthorn K, Ongaiyooth L, Vanavanan S, Sirivongs D, Thirakhupt P, Mittal B, Singh AK; Thai-SEEK Group. Prevalence and risk factors of chronic kidney disease in the Thai adult population: Thai SEEK study. Nephrol Dial Transplant. 2010 May;25(5):1567-75. doi: 10.1093/ndt/gfp669. Epub 2009 Dec 27. PMID 20037182
- See also: Research Subcommite — http://nephrothai.org